CLINICAL TRIAL: NCT03413371
Title: Influence of SPI-guided Analgesia With Preventive Different Peribulbar Blocks (PBB) on the Presence of OCR, Postoperative Pain, PONV in Patients Undergoing VRS Under General Anaesthesia: a Randomised, Controlled Trial
Brief Title: Different Peribulbar Blocks With SPI-guided Anaesthesia for VRS (P&MSPIVRS)
Acronym: PBBVRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Silesia (Other)
Collaborators: Silesian University of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SilesianMUKOAiIT8
Record Dates: First submitted 2017-12-27; First posted 2018-01-29 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2020-06

CONDITIONS: Vitreoretinal Surgeries; Postoperative Nausea and Vomiting; Postoperative Pain; Oculocardiac Reflex
Keywords: Surgical Pleth Index (SPI); General Anaesthesia (GA),; Numerical Rating Scale (NRS); Adequacy of Anaesthesia (AoA); Peribulbar Block (PBB); bupivacaine; ropivacaine; lidocaine
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Acetaminophen; Lidocaine; Bupivacaine; Ropivacaine

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Single (Participant)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0,5 % bupivacaine with of 2% lidocaine (Experimental): in group BL patients in group BF will receive regional peribulbar block using a solution of 0,5% bupivacaine (2,5 ml) with 2% lidocaine (2,5 ml)
  Interventions: Drug: paracetamol; Drug: 1 % Ropivacaine; Drug: 0,5 % bupivacaine
- 0,5 % bupivacaine (Experimental): in group B patients in group BF will receive regional peribulbar block using a solution of 0,5% bupivacaine (5 ml)
  Interventions: Drug: paracetamol; Drug: 0,5 % bupivacaine with of 2% lidocaine; Drug: 1 % Ropivacaine
- 1 % ropivacaine (Experimental): in group RL patients in group BF will receive regional peribulbar block using a solution of 1% ropivacaine (5 ml)
  Interventions: Drug: paracetamol; Drug: 0,5 % bupivacaine with of 2% lidocaine; Drug: 0,5 % bupivacaine
- paracetamol (Experimental): in P group patients will receive preemptive analgesia using 1 gram of paracetamol before induction of general anaesthesia
  Interventions: Drug: 0,5 % bupivacaine with of 2% lidocaine; Drug: 1 % Ropivacaine; Drug: 0,5 % bupivacaine

INTERVENTIONS:
Drug: paracetamol — in group P patients will receive pre-emptive analgesia using intravenous infusion of acetaminophen in a single dose of 10-15 mg per kg of body weight
  Arms: 0,5 % bupivacaine; 0,5 % bupivacaine with of 2% lidocaine; 1 % ropivacaine
Drug: 0,5 % bupivacaine with of 2% lidocaine — in group BL patients will receive regional peribulbar block using a solution of 0,5% bupivacaine (2,5 ml) with 2% lidocaine (2,5 ml)
  Other Names: Bupivacaine; Lidocaine
  Arms: 0,5 % bupivacaine; 1 % ropivacaine; paracetamol
Drug: 1 % Ropivacaine — in group R patients will receive regional peribulbar block using a solution of 0,75 % ropivacaine (5 ml)
  Other Names: ropivacaine
  Arms: 0,5 % bupivacaine; 0,5 % bupivacaine with of 2% lidocaine; paracetamol
Drug: 0,5 % bupivacaine — in group B patients will receive regional peribulbar block using a solution of 0,5% bupivacaine (5 ml)
  Other Names: bupivacaine
  Arms: 0,5 % bupivacaine with of 2% lidocaine; 1 % ropivacaine; paracetamol

SUMMARY:
The aim of this randomized trial is to assess the efficacy of preventive analgesia using different peribulbar blocks (PBB) under SPI-guided anaesthesia for vitreoretinal surgery (VRS), presence of PONV (postoperative nausea and vomiting) and oculocardiac reflex (OCR) and compare Numerical Rating Scale (NRS) with Surgical Pleth Index (SPI) for monitoring pain perception postoperatively.

Patients will receive general anaesthesia combined with either preventive PBB using either lidocaine with bupivacaine or bupivacaine or ropivacaine

DETAILED DESCRIPTION:
Monitoring depth of anaesthesia using spectral entropy (SE) and quality of neuromuscular block are routine in modern anaesthesia, whereas monitoring of analgesia still requires further studies. Recently, the Surgical Pleth Index (SPI) was added as a surrogate variable showing the nociception-antinociception balance into abovementioned parameters constituting a novel approach in monitoring patients intraoperatively, known as adequacy of anaesthesia (AoA) or tailor-made anaesthesia.

Different options of local anesthetic mixtures used for peribulbar block result in different analgetic potency. PBB is supposed to reduce requirement for intraoperative narcotic analgesics when used together with general anaesthesia and therefore may reduce the rate of PONV, OCR and perception of postoperative pain.

The aim of the study is to investigate the influence of different PBBs on abovementioned outcomes.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate in the study written consent to undergo general anaesthesia alone or combined with different techniques of pre-emptive analgesia and vitreoretinal surgery

Exclusion Criteria:

* history of allergy to local anaesthetics or paracetamol necessity of administration of vasoactive drugs influencing SPI monitoring pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
pain perception intraoperatively | intraoperative assessment
  The investigators will compare the efficacy of analgesia intraoperatively according to technique of analgesia used preoperatively: either peribulbar block or intravenous infusion. The investigators will administer a rescue dose of fentanyl intravenously in a dose of 1 mcg per kg of body weight in the case when SPI (surgical pleh index value) value increases over 15 points in SPI scale every 5 minutes until SPI value decreases back to baseline value. Additionally, the investigators will analyse rescue fentanyl consumption in abovementioned groups

SECONDARY OUTCOMES:
oculocardiac reflex rate | intraoperative assessment
  the investigators will compare the rate of presence of OCR intraoperatively in studied groups observing the presence of heart rate (HR) rapid decrease by 30%.
pain perception postoperatively | up to one hour after discharge to postoperative unit performed every 10 minutes.
  The investigators will compare the efficacy of analgesia postoperatively according to technique of analgesia used preoperatively: sort of anaesthetic mixture used for peribulbar block. The investigators will use the numeric rating scale (NRS) and compare it with surgical pleth index value (SPI) for certain pain perception: mild, moderate, acute.
PONV (postoperative nausea and vomiting) | postoperative assessment up to 24 hours
  The investigators will compare the presence of every incident of PONV after emergence from GA in studied groups and use predictive Apfel Score

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Silesia, Sosnowiec, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF
Time Frame: article in Anesthesiology and Intensive Therapy in 2021, case reports

REFERENCES:
- [Result] Gruenewald M, Herz J, Schoenherr T, Thee C, Steinfath M, Bein B. Measurement of the nociceptive balance by Analgesia Nociception Index and Surgical Pleth Index during sevoflurane-remifentanil anesthesia. Minerva Anestesiol. 2015 May;81(5):480-9. Epub 2014 Jul 17. PMID 25032676
- [Result] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Result] Gruenewald M, Ilies C. Monitoring the nociception-anti-nociception balance. Best Pract Res Clin Anaesthesiol. 2013 Jun;27(2):235-47. doi: 10.1016/j.bpa.2013.06.007. PMID 24012235
- [Result] Gruenewald M, Willms S, Broch O, Kott M, Steinfath M, Bein B. Sufentanil administration guided by surgical pleth index vs standard practice during sevoflurane anaesthesia: a randomized controlled pilot study. Br J Anaesth. 2014 May;112(5):898-905. doi: 10.1093/bja/aet485. Epub 2014 Feb 16. PMID 24535604
- [Result] Jaichandran VV, Raman R, Gella L, Sharma T. Local anesthetic agents for vitreoretinal surgery: no advantage to mixing solutions. Ophthalmology. 2015 May;122(5):1030-3. doi: 10.1016/j.ophtha.2014.11.026. Epub 2015 Jan 10. PMID 25582785
- [Result] Ghali AM. The efficacy of 0.75% levobupivacaine versus 0.75% ropivacaine for peribulbar anesthesia in vitreoretinal surgery. Saudi J Anaesth. 2012 Jan;6(1):22-6. doi: 10.4103/1658-354X.93050. PMID 22412772
- [Result] Seidenari P, Santin G, Milani P, David A. Peribulbar and retrobulbar combined anesthesia for vitreoretinal surgery using ropivacaine. Eur J Ophthalmol. 2006 Mar-Apr;16(2):295-9. doi: 10.1177/112067210601600216. PMID 16703549
- [Result] Subramaniam R, Subbarayudu S, Rewari V, Singh RP, Madan R. Usefulness of pre-emptive peribulbar block in pediatric vitreoretinal surgery: a prospective study. Reg Anesth Pain Med. 2003 Jan-Feb;28(1):43-7. doi: 10.1053/rapm.2003.50032. PMID 12567343
- [Result] Fekrat S, Elsing SH, Raja SC, Campochiaro PA, de Juan E Jr, Haller JA. Eye pain after vitreoretinal surgery: a prospective study of 185 patients. Retina. 2001;21(6):627-32. doi: 10.1097/00006982-200112000-00010. PMID 11756886
- [Result] Calenda E, Olle P, Muraine M, Brasseur G. Peribulbar anesthesia and sub-Tenon injection for vitreoretinal surgery: 300 cases. Acta Ophthalmol Scand. 2000 Apr;78(2):196-9. doi: 10.1034/j.1600-0420.2000.078002196.x. PMID 10794256
- [Result] Sajedi P, Nejad MS, Montazeri K, Baloochestani E. Comparing the preventive effect of 2 percent topical lidocaine and intravenous atropine on oculocardiac reflex in ophthalmological surgeries under general anesthesia. Int J Prev Med. 2013 Nov;4(11):1258-65. PMID 24404359
- [Result] Calenda E, Quintyn JC, Brasseur G. Peribulbar anaesthesia using a combination of lidocaine, bupivocaine and clonidine in vitreoretinal surgery. Indian J Ophthalmol. 2002 Sep;50(3):205-8. PMID 12355695
- [Result] Mandelcorn M, Taback N, Mandelcorn E, Ananthanarayan C. Risk factors for pain and nausea following retinal and vitreous surgery under conscious sedation. Can J Ophthalmol. 1999 Aug;34(5):281-5. PMID 10486687